CLINICAL TRIAL: NCT05536440
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR OPEN, PLACEBO CONTROLLED, DOSE ESCALATING STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND PHARMACODYNAMICS OF SINGLE INTRAVENOUS AND MULTIPLE SUBCUTANEOUS AND INTRAVENOUS DOSES OF PF-07261271 IN HEALTHY PARTICIPANTS
Brief Title: A Study to Learn About Study Medicine Called PF-07261271 in Healthy People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: C4631001
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: Healthy volunteer; Healthy; IBD; Inflammatory bowel disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (16):
- Cohort 1 active (Experimental): Dose A
  Interventions: Drug: PF-07261271
- Cohort 1 placebo (Placebo Comparator): Dose A
  Interventions: Drug: Placebo
- Cohort 2 active (Experimental): Dose B
  Interventions: Drug: PF-07261271
- Cohort 2 placebo (Placebo Comparator): Dose B
  Interventions: Drug: Placebo
- Cohort 3 active (Experimental): Dose C
  Interventions: Drug: PF-07261271
- Cohort 3 placebo (Placebo Comparator): Dose C
  Interventions: Drug: Placebo
- Cohort 4 active (Experimental): Dose D
  Interventions: Drug: PF-07261271
- Cohort 4 placebo (Placebo Comparator): Dose D
  Interventions: Drug: Placebo
- Cohort 5 active (Experimental): Dose E
  Interventions: Drug: PF-07261271
- Cohort 5 placebo (Placebo Comparator): Dose E
  Interventions: Drug: Placebo
- Cohort 6 active (Experimental): Dose F
  Interventions: Drug: PF-07261271
- Cohort 6 placebo (Placebo Comparator): Dose F
  Interventions: Drug: Placebo
- Cohort 7 active (Experimental): Dose G
  Interventions: Drug: PF-07261271
- Cohort 7 placebo (Placebo Comparator): Dose G
  Interventions: Drug: Placebo
- Cohort 8 active (Experimental): Dose H
  Interventions: Drug: PF-07261271
- Cohort 8 placebo (Placebo Comparator): Dose H
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-07261271 — IV or SC
  Arms: Cohort 1 active; Cohort 2 active; Cohort 3 active; Cohort 4 active; Cohort 5 active; Cohort 6 active; Cohort 7 active; Cohort 8 active
Drug: Placebo — IV or SC
  Arms: Cohort 1 placebo; Cohort 2 placebo; Cohort 3 placebo; Cohort 4 placebo; Cohort 5 placebo; Cohort 6 placebo; Cohort 7 placebo; Cohort 8 placebo

SUMMARY:
The purpose of this clinical trial is to learn about the safety and effects of the study medicine PF-07261271 for the potential treatment of Inflammatory Bowel Disease.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals as determined by medical evaluation
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

* Clinically significant medical conditions
* History of HIV infection, hepatitis B, or hepatitis C
* BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic)
* Clinically relevant ECG abnormalities
* Previous study drug administration within 30 days or 5 half-lives of first planned dose
* History of drug/alcohol abuse or >20 cigarettes/day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Orange County Research Center, Lake Forest, California
  - Orange County Research Center, Tustin, California
  - Clinilabs, Eatontown, New Jersey
  - ICON, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4631001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 35 participants (27 participants assigned to single ascending dose [SAD] cohorts and 8 participants assigned in the multiple doses [MD] cohorts) were enrolled in the study.
Pre-assignment Details: In this study, dose have been reported from dose levels 1 to 4, wherein dose level 1 is the lowest dose and dose level 4 is the highest dose received by the study participants.
Groups:
- SAD: Placebo: Healthy participants who were randomized to receive placebo matched to PF-07261271 as single intravenous (IV) dose on Day 1.
- SAD: PF-07261271 Dose Level 1: Healthy participants who were randomized to receive PF-07261271 Dose Level 1 as single IV dose on Day 1.
- SAD: PF-07261271 Dose Level 2: Healthy participants who were randomized to receive PF-07261271 Dose Level 2 as single IV dose on Day 1.
- SAD: PF-07261271 Dose Level 3: Healthy participants who were randomized to receive PF-07261271 Dose Level 3 as single IV dose on Day 1.
- SAD: PF-07261271 Dose Level 4: Healthy participants who were randomized to receive PF-07261271 Dose Level 4 as single IV dose on Day 1.
- SAD: Placebo (Japanese Participants): Healthy Japanese participants who were randomized to receive placebo matched to PF-07261271 as single dose on Day 1.
- SAD: PF-07261271 Dose Level 4 (Japanese Participants): Healthy Japanese participants who were randomized to receive PF-07261271 Dose Level 4 as single IV dose on Day 1.
- MD: Placebo: Healthy participants who were randomized to receive placebo matched to PF-07261271 as repeated subcutaneous (SC) doses on Day 1 and Day 29.
- MD: PF-07261271 Dose Level 3: Healthy participants who were randomized to receive PF-07261271 Dose Level 3 repeated SC doses on Day 1 and Day 29.
Period: Overall Study
Arm/Group | SAD: Placebo | SAD: PF-07261271 Dose Level 1 | SAD: PF-07261271 Dose Level 2 | SAD: PF-07261271 Dose Level 3 | SAD: PF-07261271 Dose Level 4 | SAD: Placebo (Japanese Participants) | SAD: PF-07261271 Dose Level 4 (Japanese Participants) | MD: Placebo | MD: PF-07261271 Dose Level 3
Started | 8 | 2 | 2 | 4 | 6 | 1 | 4 | 2 | 6
Completed | 8 | 2 | 2 | 4 | 6 | 1 | 4 | 2 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- SAD: Placebo: Healthy participants who were randomized to receive placebo matched to PF-07261271 as single IV dose on Day 1.
- MD: PF-07261271 Dose Level 3: Healthy participants who were randomized to receive PF-07261271 Dose level 3 repeated escalating SC doses on Day 1 and Day 29.
- Total: Total of all reporting groups
Arm/Group | SAD: Placebo | SAD: PF-07261271 Dose Level 1 | SAD: PF-07261271 Dose Level 2 | SAD: PF-07261271 Dose Level 3 | SAD: PF-07261271 Dose Level 4 | SAD: Placebo (Japanese Participants) | SAD: PF-07261271 Dose Level 4 (Japanese Participants) | MD: Placebo | MD: PF-07261271 Dose Level 3 | Total
Number analyzed (Participants) | 8 | 2 | 2 | 4 | 6 | 1 | 4 | 2 | 6 | 35
Age, Customized [Count of Participants; unit: Participants]
  Less than (<) 18 Years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18-25 Years | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  26-35 Years | 2 | 1 | 2 | 2 | 1 | 0 | 0 | 1 | 3 | 12
  36-45 Years | 2 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 6
  Greater than (>) 45 Years | 2 | 0 | 0 | 2 | 2 | 1 | 3 | 1 | 3 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 10
  Male | 5 | 1 | 2 | 3 | 5 | 1 | 3 | 1 | 4 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 6
  Not Hispanic or Latino | 6 | 2 | 1 | 4 | 4 | 1 | 4 | 2 | 5 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 5
  White | 6 | 2 | 1 | 4 | 3 | 0 | 0 | 1 | 6 | 23
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs): SAD Cohort
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE was considered a TEAE if the event started during the effective duration of treatment. All events that started on or after the first dosing day and time/start time, if collected, but before the end of the last follow-up date, were considered as TEAEs. AEs included all SAEs and Non-SAEs.
Time Frame: From start of study intervention (Day 1) up to end of study, approximately up to 15 months
Population: Safety analysis set included all participants randomly assigned to study intervention who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- SAD: Placebo (Japanese Participants): Healthy Japanese participants who were randomized to receive placebo matched to PF-07261271 as single IV dose on Day 1.
Arm/Group | SAD: Placebo | SAD: PF-07261271 Dose Level 1 | SAD: PF-07261271 Dose Level 2 | SAD: PF-07261271 Dose Level 3 | SAD: PF-07261271 Dose Level 4 | SAD: Placebo (Japanese Participants) | SAD: PF-07261271 Dose Level 4 (Japanese Participants)
Number analyzed (Participants) | 8 | 2 | 2 | 4 | 6 | 1 | 4
Participants | 4 | 1 | 1 | 3 | 2 | 0 | 1

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs): MD Cohort
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE was considered a TEAE if the event started during the effective duration of treatment. All events that started on or after the first dosing day and time/start time, if collected, but before the end of the last follow-up date, were considered as TEAEs. AEs included all SAEs and Non-SAEs.
Time Frame: From start of study intervention (Day 1) up to end of study, approximately of 15.5 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- MD: Placebo: Healthy participants who were randomized to receive placebo matched to PF-07261271 as repeated SC doses on Day 1 and Day 29.
Arm/Group | MD: Placebo | MD: PF-07261271 Dose Level 3
Number analyzed (Participants) | 2 | 6
Participants | 2 | 5

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs): SAD Cohort
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. SAEs were defined as any untoward medical occurrence that, at any dose, met one or more of the criteria: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic or other medically significant event.
Time Frame: From start of study intervention (Day 1) up to end of study, approximately up to 15 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SAD: Placebo | SAD: PF-07261271 Dose Level 1 | SAD: PF-07261271 Dose Level 2 | SAD: PF-07261271 Dose Level 3 | SAD: PF-07261271 Dose Level 4 | SAD: Placebo (Japanese Participants) | SAD: PF-07261271 Dose Level 4 (Japanese Participants)
Number analyzed (Participants) | 8 | 2 | 2 | 4 | 6 | 1 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs): MD Cohort
Description: as for outcome 3
Time Frame: From start of study intervention (Day 1) up to end of study, approximately of 15.5 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MD: Placebo | MD: PF-07261271 Dose Level 3
Number analyzed (Participants) | 2 | 6
Participants | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs Abnormalities: SAD Cohort
Description: Criteria for abnormal values of vital signs: systolic blood pressure (millimeters of mercury [mmHg]) value less than (<) 90 mmHg, change greater than or equal to (>=) 30 mmHg increase, change >= 30 mmHg decrease; diastolic blood pressure (mmHg), value <50 mmHg, change >=20 mmHg increase, change >=20 mmHg decrease; pulse rate (beats per minute [bpm]) value <40bpm, value greater than (>) 120bpm. Clinical significance was determined based on investigator's discretion.
Time Frame: From start of study intervention (Day 1) up to end of study, approximately up to 15 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SAD: Placebo | SAD: PF-07261271 Dose Level 1 | SAD: PF-07261271 Dose Level 2 | SAD: PF-07261271 Dose Level 3 | SAD: PF-07261271 Dose Level 4 | SAD: Placebo (Japanese Participants) | SAD: PF-07261271 Dose Level 4 (Japanese Participants)
Number analyzed (Participants) | 8 | 2 | 2 | 4 | 6 | 1 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs Abnormalities: MD Cohort
Description: Criteria for abnormal values of vital signs: systolic blood pressure (mmHg) value < 90 mmHg, change >= 30 mmHg increase, change >= 30 mmHg decrease; diastolic blood pressure (mmHg), value <50 mmHg, change >=20 mmHg increase, change >=20 mmHg decrease; pulse rate (bpm) value < 40bpm, value > 120bpm. Clinical significance was determined based on investigator's discretion.
Time Frame: From start of study intervention (Day 1) up to end of study, approximately of 15.5 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MD: Placebo | MD: PF-07261271 Dose Level 3
Number analyzed (Participants) | 2 | 6
Participants | 0 | 0

7. Primary Outcome: Number of Participants With Clinically Significant Changes in Laboratory Abnormalities: SAD Cohort
Description: Criteria:Hematology(Activated partial thromboplastin time>1.1*upper limit of normal(ULN); Basophils &eosinophils>1.2*ULN; erythrocytes,hematocrit,hemoglobin,lymphocytes,neutrophils <0.8*lower limit of normal(LLN); leukocytes <0.6*LLN, >1.5*ULN; monocytes >1.2*ULN; platelets <0.5*LLN; prothrombin international randomized ratio &prothrombin Time >1.1*ULN), clinical chemistry (alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase >3.0*ULN; albumin, protein <0.8*LLN, >1.2*ULN; bicarbonate, calcium, chloride, potassium <0.9*LLN,>1.1*ULN; bilirubin >1.5*ULN; creatinine >1.3*ULN; glucose, Glucose-FASTING <0.6*LLN,>1.5*ULN; Sodium <0.95*LLN,>1.05*ULN; Urate: >1.2*ULN;Urea Nitrogen: >1.3*ULN),urinalysis(Bacteria > 20;epithelial cells >=6;granular, hyaline, RBC&WBC casts >1;ketones,leukocyte esterase, nitrite, urine glucose, urine hemoglobin, urine protein>=1,urine erythrocytes,leukocytes >=20;pH(scalar)<4.5,>8.Clinical significance determined on investigator's discretion.
Time Frame: From start of study intervention (Day 1) up to end of study, approximately up to 15 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SAD: Placebo | SAD: PF-07261271 Dose Level 1 | SAD: PF-07261271 Dose Level 2 | SAD: PF-07261271 Dose Level 3 | SAD: PF-07261271 Dose Level 4 | SAD: Placebo (Japanese Participants) | SAD: PF-07261271 Dose Level 4 (Japanese Participants)
Number analyzed (Participants) | 8 | 2 | 2 | 4 | 6 | 1 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Clinically Significant Changes in Laboratory Abnormalities: MD Cohort
Description: as for outcome 7
Time Frame: From start of study intervention (Day 1) up to end of study, approximately of 15.5 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MD: Placebo | MD: PF-07261271 Dose Level 3
Number analyzed (Participants) | 2 | 6
Participants | 0 | 0

9. Primary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Abnormalities: SAD Cohort
Description: Criteria for abnormal values of ECG parameters: pulse rate (PR) interval greater than or equal to (>=)300 milliseconds (msec); PR interval change >=25 percent (%) or >=50 %, QRS interval >=140 msec and QRS interval change: >=50%. QT interval using Fridericia's correction (QTcF) range from 450 msec to less than (<)480 msec, less than (<) 480 msec to maximum less than or equal to (<=)500 msec, >500 msec, <=30 to <60 msec and >=60 msec. Only rows which included at least 1 participant with abnormality are reported in this outcome measure. Clinical significance was determined based on investigator's discretion.
Time Frame: From start of study intervention (Day 1) up to end of study, approximately up to 15 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SAD: Placebo | SAD: PF-07261271 Dose Level 1 | SAD: PF-07261271 Dose Level 2 | SAD: PF-07261271 Dose Level 3 | SAD: PF-07261271 Dose Level 4 | SAD: Placebo (Japanese Participants) | SAD: PF-07261271 Dose Level 4 (Japanese Participants)
Number analyzed (Participants) | 8 | 2 | 2 | 4 | 6 | 1 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Clinically Significant Changes in ECG Abnormalities: MD Cohort
Description: as for outcome 9
Time Frame: From start of study intervention (Day 1) up to end of study, approximately of 15.5 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MD: Placebo | MD: PF-07261271 Dose Level 3
Number analyzed (Participants) | 2 | 6
Participants | 0 | 0

11. Secondary Outcome: Area Under the Concentration Versus Time Curve From Time Zero to the Last Quantifiable Time Point (AUClast) of PF-07261271: SAD Cohort
Description: AUClast was determined using Linear Log trapezoidal method.
Time Frame: Predose and 0, 2, 4, 8, 12, 24, 48, 72, 192, 360, 768, 1104, 1464, 2184, 4344, 5064, 5784, 6504, 7224, 7944, 8664, 10824 hours post dose
Population: Pharmacokinetic (PK) parameter analysis population included all randomized participants who received at least 1 dose of PF-07261271 and who had at least 1 of the PK parameters of interest calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms*hour per milliliter
Arm/Group | SAD: PF-07261271 Dose Level 1 | SAD: PF-07261271 Dose Level 2 | SAD: PF-07261271 Dose Level 3 | SAD: PF-07261271 Dose Level 4 | SAD: PF-07261271 Dose Level 4 (Japanese Participants)
Number analyzed (Participants) | 2 | 2 | 4 | 6 | 4
Nanograms*hour per milliliter | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 3740000 Nanograms*hour per milliliter (ng*hr/mL) and 4200000 ng*hr/mL. | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 16300000 ng*hr/mL and 20000000 ng*hr/mL. | 65600000 (35) | 324100000 (18) | 345000000 (28)

12. Secondary Outcome: Area Under the Serum Concentration Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of PF-07261271: SAD Cohort
Description: AUCinf was determined as AUClast + (Clast*/kel), where Clast* is the predicted serum concentration at the last quantifiable time point estimated from the log-linear regression analysis.
Time Frame: as for outcome 11
Population: PK parameter analysis population included all randomized participants who received at least 1 dose of PF-07261271 and who had at least 1 of the PK parameters of interest calculated. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms*hour per milliliter
Arm/Group | SAD: PF-07261271 Dose Level 1 | SAD: PF-07261271 Dose Level 2 | SAD: PF-07261271 Dose Level 3 | SAD: PF-07261271 Dose Level 4 | SAD: PF-07261271 Dose Level 4 (Japanese Participants)
Number analyzed (Participants) | 2 | 2 | 3 | 6 | 4
Nanograms*hour per milliliter | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 3740000 ng*hr/mL and 4530000 ng*hr/mL. | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 16600000 ng*hr/mL and 21300000 ng*hr/mL. | 61010000 (36) | 332600000 (18) | 368100000 (28)

13. Secondary Outcome: Maximum Plasma Concentration (Cmax) of PF-07261271: SAD Cohort
Description: Cmax was defined as maximum serum concentration.
Time Frame: as for outcome 11
Population: PK parameter analysis population included all randomized participants who received at least 1 dose of PF-07261271 and who had at least 1 of the PK parameters of interest calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | SAD: PF-07261271 Dose Level 1 | SAD: PF-07261271 Dose Level 2 | SAD: PF-07261271 Dose Level 3 | SAD: PF-07261271 Dose Level 4 | SAD: PF-07261271 Dose Level 4 (Japanese Participants)
Number analyzed (Participants) | 2 | 2 | 4 | 6 | 4
Nanograms per milliliter | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 10400 ng/mL and 10500 ng/mL. | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 46900 ng/mL and 50000 ng/mL. | 143300 (21) | 372800 (17) | 313900 (31)

14. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of PF-07261271: SAD Cohort
Description: Tmax was defined as time for Cmax.
Time Frame: as for outcome 11
Population: as for outcome 13
Measure: Median (Full Range); unit: Hours
Arm/Group | SAD: PF-07261271 Dose Level 1 | SAD: PF-07261271 Dose Level 2 | SAD: PF-07261271 Dose Level 3 | SAD: PF-07261271 Dose Level 4 | SAD: PF-07261271 Dose Level 4 (Japanese Participants)
Number analyzed (Participants) | 2 | 2 | 4 | 6 | 4
Hours | NA [NA to NA] — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 2.00 hours and 2.00 hours. | NA [NA to NA] — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 1.08 hours and 13.2 hours. | 2.12 [1.00 to 4.00] | 3.13 [0.967 to 5.53] | 5.26 [2.17 to 48.0]

15. Secondary Outcome: Terminal Elimination Half-life (t1/2) of PF-07261271: SAD Cohort
Description: t1/2 was determined using Loge (2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log linear -concentration time- curve.
Time Frame: as for outcome 11
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | SAD: PF-07261271 Dose Level 1 | SAD: PF-07261271 Dose Level 2 | SAD: PF-07261271 Dose Level 3 | SAD: PF-07261271 Dose Level 4 | SAD: PF-07261271 Dose Level 4 (Japanese Participants)
Number analyzed (Participants) | 2 | 2 | 3 | 6 | 4
Hours | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 158 hours and 328 hours. | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 297 hours and 299 hours. | 330.7 (193.29) | 1533 (324.39) | 1529 (1018.5)

16. Secondary Outcome: Area Under the Concentration Time Profile From Time Zero to Time Tau (τ), the Dosing Interval (AUCtau) of PF-07261271: MD Cohort
Description: AUCtau was defined as area under the concentration time profile from time zero to time tau (τ), the dosing interval, where tau=672 hours for every 4-week dosing. AUCtau was determined by Linear Log trapezoidal method.
Time Frame: Predose and 0, 2, 4, 8, 12, 48, 96, 192, 360, 720, 744, 1224, 1584, 1944, 2664, 4104, 4824, 5544, 6264, 6984, 7704, 8424, 9144 and 11304 hours post-dose on Day 1 and 29
Population: PK parameter analysis population included all randomized participants who received at least 1 dose of PF-07261271 and who had at least 1 of the PK parameters of interest calculated. Here, 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms*hour per milliliter
Arm/Group | MD: PF-07261271 Dose Level 3
Number analyzed (Participants) | 6
Nanograms*hour per milliliter
  Day 1 | 17600000 (27)
  Day 29: number analyzed (Participants) | 5
  Day 29 | 27900000 (22)

17. Secondary Outcome: Cmax of PF-07261271: MD Cohort
Description: Cmax was defined as maximum serum concentration.
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms*hour per milliliter
Arm/Group | MD: PF-07261271 Dose Level 3
Number analyzed (Participants) | 6
Nanograms*hour per milliliter
  Day 1 | 34120 (28)
  Day 29: number analyzed (Participants) | 5
  Day 29 | 49600 (28)

18. Secondary Outcome: Tmax of PF-07261271: MD Cohort
Description: Tmax was defined as time for Cmax.
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Median (Full Range); unit: Hours
Arm/Group | MD: PF-07261271 Dose Level 3
Number analyzed (Participants) | 6
Hours
  Day 1 | 253 [48.0 to 338]
  Day 29: number analyzed (Participants) | 5
  Day 29 | 170 [48.0 to 172]

19. Secondary Outcome: Terminal Elimination Half-life (t1/2) of PF-07261271: MD Cohort
Description: as for outcome 15
Time Frame: as for outcome 16
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | MD: PF-07261271 Dose Level 3
Number analyzed (Participants) | 6
Hours | 1150 (856.40)

20. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) Against PF-07261271: SAD Cohort
Description: ADA positive was defined as ADA titer >= 100; ADA negative defined as ADA titer < 100. Baseline was defined as the last pre-dose measurement
Time Frame: Baseline up to 15 months
Population: Immunogenicity data analysis was performed on the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD: PF-07261271 Dose Level 1 | SAD: PF-07261271 Dose Level 2 | SAD: PF-07261271 Dose Level 3 | SAD: PF-07261271 Dose Level 4 | SAD: PF-07261271 Dose Level 4 (Japanese Participants)
Number analyzed (Participants) | 2 | 2 | 4 | 6 | 4
Participants | 2 | 2 | 4 [lower limit 19690.28] | 6 | 4

21. Secondary Outcome: Number of Participants With ADA Against PF-07261271: MD Cohort
Description: ADA positive defined as ADA titer >= 100; ADA negative defined as ADA titer < 100. Baseline was defined as the last pre-dose measurement.
Time Frame: Baseline up to 15.5 months
Population: Immunogenicity data analysis was performed on the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | MD: PF-07261271 Dose Level 3
Number analyzed (Participants) | 6
Participants | 6 [lower limit 32249.01]

22. Secondary Outcome: Number of Participants With Neutralizing Antibodies (NAb) Against PF-07261271: SAD Cohort
Description: NAb was determined by electrochemiluminescent (ECL) competitive ligand binding assay using the Meso Scale Discovery (MSD) platform.
Time Frame: Baseline up to 15 months
Population: Immunogenicity data analysis was performed on the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD: PF-07261271 Dose Level 1 | SAD: PF-07261271 Dose Level 2 | SAD: PF-07261271 Dose Level 3 | SAD: PF-07261271 Dose Level 4 | SAD: PF-07261271 Dose Level 4 (Japanese Participants)
Number analyzed (Participants) | 2 | 2 | 4 | 6 | 4
Participants | 2 | 2 | 4 [lower limit 19690.28] | 5 | 2

23. Secondary Outcome: Number of Participants With NAb Against PF-07261271: MD Cohort
Description: as for outcome 22
Time Frame: Baseline up to 15.5 months
Population: Immunogenicity data analysis was performed on the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | MD: PF-07261271 Dose Level 3
Number analyzed (Participants) | 6
Participants | 5 [lower limit 32249.01]

ADVERSE EVENTS:
Time Frame: SAD Cohort: From start of study intervention (Day 1) up to approximately 15 months and MD Cohort: From start of study intervention (Day 1) up to approximately 15.5 months
Description: Safety analysis set included all participants randomly assigned to study intervention who took at least 1 dose of study intervention.
Groups:
- MD: Placebo: Healthy participants who were randomized to receive placebo matched to PF-07261271 as repeated SC dose on Day 1 and Day 29.
- MD: PF-07261271 Dose Level 3: Healthy participants who were randomized to receive PF-07261271 300 mg repeated escalating SC doses on Day 1 and Day 29.
Arm/Group | SAD: Placebo | SAD: PF-07261271 Dose Level 1 | SAD: PF-07261271 Dose Level 2 | SAD: PF-07261271 Dose Level 3 | SAD: PF-07261271 Dose Level 4 | SAD: Placebo (Japanese Participants) | SAD: PF-07261271 Dose Level 4 (Japanese Participants) | MD: Placebo | MD: PF-07261271 Dose Level 3
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/2 | 0/2 | 0/4 | 0/6 | 0/1 | 0/4 | 0/2 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/2 | 0/2 | 0/4 | 0/6 | 0/1 | 0/4 | 0/2 | 0/6
Other Adverse Events (participants affected / at risk) | 4/8 | 1/2 | 1/2 | 3/4 | 2/6 | 0/1 | 1/4 | 2/2 | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SAD: Placebo (N=8) | SAD: PF-07261271 Dose Level 1 (N=2) | SAD: PF-07261271 Dose Level 2 (N=2) | SAD: PF-07261271 Dose Level 3 (N=4) | SAD: PF-07261271 Dose Level 4 (N=6) | SAD: Placebo (Japanese Participants) (N=1) | SAD: PF-07261271 Dose Level 4 (Japanese Participants) (N=4) | MD: Placebo (N=2) | MD: PF-07261271 Dose Level 3 (N=6)
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT05536440/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT05536440/SAP_001.pdf